CLINICAL TRIAL: NCT03606369
Title: Effectiveness and Quality of Life Analysis of Palonosetron Against Ondansetron Combined With Dexamethasone and Fosaprepitant in Prevention of Acute and Delayed Emesis Associated to Chemotherapy Moderate and Highly Emetogenic in Breast Cancer.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Responsible Party: Principal Investigator, Claudia Arce-Salinas, Attendin physician, Instituto Nacional de Cancerologia de Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CE1002/15
Record Dates: First submitted 2018-07-03; First posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Breast Neoplasm; Antineoplastic Agents; Antiemetics; Quality of Life
Keywords: Breast Neoplasm; Antiemetics; Quality of Life; Palonosetron; Ondansetron
MeSH Terms: conditions — Breast Neoplasms | interventions — Palonosetron; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Palonosetron (Experimental): Early emesis: Palonosetron 0.25 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV.
  Delayed emesis: Dexamethasone 8 mg orally on days 2, 3 and 4.
  Interventions: Drug: Palonosetron
- Ondansetron (Active Comparator): Early emesis: Ondansetron 16 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV.
  Delayed emesis: Metoclopramide 10 mg orally every 6 hours + Dexamethasone 8 mg orally every 24 hrs.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Palonosetron — Palonosetron 0.25 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV for early emesis and for delayed emesis Dexamethasone 8 mg orally on days 2, 3 and 4.
  Arms: Palonosetron
Drug: Ondansetron — Early emesis: Ondansetron 16 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV. and for delayed emesis: Metoclopramide 10 mg orally every 6 hours + Dexamethasone 8 mg orally every 24 hrs.
  Arms: Ondansetron

SUMMARY:
Nausea and vomiting are common complications on the chemotherapy (CT) and can affect the quality of life (QoL) of the patients. If not treated adequately it can produce other problems such as dehydration, weight loss, fatigue and even can induce the non-compliance of the treatment. In extreme cases it can put the patient ́s life at risk. There are various antiemetic treatments that vary both in cost and effectiveness. It ́s important to determine which are the strategies that are most effective and can improve the QoL of the patients.

Methodology:

The analysis will be done in patients who receive adjuvant and neoadjuvant chemotherapy and that have not received previously chemotherapy or radiotherapy, they will be stratified according to the emetogenic potential of the CT. They were given a diary of symptoms to register any discomfort suffered after receiving their treatment and also a quality of life questionnaire was applied previous to their first cycle and previous to their second cycle.

The patients were divided in two groups receiving either A scheme (palonosetron) or B scheme (ondansetron) in combination with dexamethasone and fosaprepitant for prevention of early emesis and Dexamethasone to group A or Dexamethasone + metoclopramide to group B for prevention of delayed emesis. As well It was analyzed the three most prevalent single nucleotide polymorphisms (SNPs) on gene ABCB1 using PCR.

The aim of this study is to evaluate the efficacy and quality of life provided by the 2 regimes noted above based on Mexican population so the results obtained can be applied widely in our country.

DETAILED DESCRIPTION:
Nausea and vomiting are common complications on the chemotherapy (CT) and can affect the quality of life (QoL) of the patients. If not treated adequately Nausea and vomiting can produce other problems such as dehydration, weight loss, fatigue and even can induce the non-compliance of the treatment. In extreme cases it can put the patient ́s life at risk. There are various antiemetic treatments that vary both in cost and effectiveness. It ́s important to determine which are the strategies that are most effective and can improve the QoL of the patients.

Methodology:

Effectiveness and quality of life analysis of patients with breast cancer that will receive adjuvant and neoadjuvant chemotherapy highly and moderately emetic chemotherapy (adriamycin and cyclophosphamide (AC), docetaxel and carboplatin (TC), docetaxel, carboplatin and trastuzumab (THC)); there will only be consider those patients that are candidates to receive CT for the first time and should have central venous access. There will be excluded patients that had received previously any kind of chemotherapy or radiotherapy. The follow-up will exclusively be done during the first cycle of CT. Patients will be stratified according to the emetogenic potential of the CT regimen ad not by the clinical stage or the histologic type of the tumor.

To keep a follow-up of the patient there will be provided symptomatic diaries where the patient can register any discomfort suffered after receiving their treatment. Along with this, there will be applied quality of life questionnaires, one previous to the CT and one previous to the second cycle.

There a proposed two regimes on antiemetic treatment. The randomization is as follows.

Group A Early emesis: Palonosetron 0.25 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV Delayed emesis: Dexamethasone 8 mg orally on days 2, 3 and 4.

Group B Early Emesis: Ondansetron 16 mg IV + Dexamethasone 12 mg IV + Fosaprepitant 150 mg IV Delayed Emesis: Metoclopramide 10 mg orally every 6 hours + Dexamethasone 8 mg orally every 24 hrs.

Considering the absence of at least one event of nausea and vomiting as a measure of effectiveness, it will be calculated the effectiveness ratio, as well as the QoL questionnaires before and after the first chemotherapy.

Finally, previously to the application of the treatment there will be obtained a peripheral blood sample for its analysis on translational medicine laboratory. There will be a process of extraction of Deoxyribonucleic Acid accordingly to the guides and the sample will be analyzed by a protein chain reaction (PCR) to detect the three most prevalent polymorphisms (SNPs)on gene ABCB1.

H0: There ́s no difference in cost - effectiveness ratio in antiemetic therapy (acute and delayed) between A and B schemes.

H1: Scheme A is superior than scheme B in 10 % for prevention of acute nausea and vomiting and 6% in delayed nausea and vomiting.

Applications:

The guides that are actually used for the antiemetic treatments are based in non Mexican populations. With this study it is expected to design an effective strategy that can be applied in mexican population

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years old or more.
* Not metastatic breast cancer confirmed with biopsy.
* Candidates to receive chemotherapy with anthracyclines combined with cyclophosphamide or carboplatin combined with docetaxel or docetaxel combined with cyclophosphamide.
* No previous treatment with radiotherapy or chemotherapy.
* Adequate hematologic function (Hb >10 gr/dl, neutrophils >1500, platelets >100,000,) renal (Creatinine <1.2 or creatinine depuration >60 ml/min), hepatic (liver enzymes <2.5 their normal value) and cardiologic (electrocardiogram).
* Adequate physical state (ECOG 0-1)
* Patients that accept to enter in protocol and sign the informed consent.

Exclusion Criteria:

* Prolonged QT (>480 mseg)
* Comorbidities of the airway
* Intolerance to swallow medications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2015-11-05 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Acute nausea control | Within the first 24 hours after first dose of chemotherapy
  Personal diary of symptoms given to the patient

SECONDARY OUTCOMES:
Delayed nausea control | Between 24 and 120 hours after first dose of chemotherapy
  Personal diary of symptoms given to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Claudia H Arce Salinas, MD, Principal Investigator
Locations (1):
- Instituto Nacional de Cancerología, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Coates A, Abraham S, Kaye SB, Sowerbutts T, Frewin C, Fox RM, Tattersall MH. On the receiving end--patient perception of the side-effects of cancer chemotherapy. Eur J Cancer Clin Oncol. 1983 Feb;19(2):203-8. doi: 10.1016/0277-5379(83)90418-2. PMID 6681766
- [Result] Craig JB, Powell BL. The management of nausea and vomiting in clinical oncology. Am J Med Sci. 1987 Jan;293(1):34-44. doi: 10.1097/00000441-198701000-00008. PMID 3544842
- [Result] Passik SD, Kirsh KL, Rosenfeld B, McDonald MV, Theobald DE. The changeable nature of patients' fears regarding chemotherapy: implications for palliative care. J Pain Symptom Manage. 2001 Feb;21(2):113-20. doi: 10.1016/s0885-3924(00)00249-9. PMID 11226762
- [Result] Hesketh PJ. Chemotherapy-induced nausea and vomiting. N Engl J Med. 2008 Jun 5;358(23):2482-94. doi: 10.1056/NEJMra0706547. No abstract available. PMID 18525044
- [Result] Grunberg SM, Warr D, Gralla RJ, Rapoport BL, Hesketh PJ, Jordan K, Espersen BT. Evaluation of new antiemetic agents and definition of antineoplastic agent emetogenicity--state of the art. Support Care Cancer. 2011 Mar;19 Suppl 1:S43-7. doi: 10.1007/s00520-010-1003-x. Epub 2010 Oct 24. PMID 20972805
- [Result] Hatoum HT, Lin SJ, Buchner D, Cox D. Comparative clinical effectiveness of various 5-HT3 RA antiemetic regimens on chemotherapy-induced nausea and vomiting associated with hospital and emergency department visits in real world practice. Support Care Cancer. 2012 May;20(5):941-9. doi: 10.1007/s00520-011-1165-1. Epub 2011 May 1. PMID 21533811
- [Result] Grunberg SM, Deuson RR, Mavros P, Geling O, Hansen M, Cruciani G, Daniele B, De Pouvourville G, Rubenstein EB, Daugaard G. Incidence of chemotherapy-induced nausea and emesis after modern antiemetics. Cancer. 2004 May 15;100(10):2261-8. doi: 10.1002/cncr.20230. PMID 15139073
- [Result] Wickham R. Evolving treatment paradigms for chemotherapy-induced nausea and vomiting. Cancer Control. 2012 Apr;19(2 Suppl):3-9. doi: 10.1177/107327481201902s02. PMID 22488022
- [Result] Schnell FM. Chemotherapy-induced nausea and vomiting: the importance of acute antiemetic control. Oncologist. 2003;8(2):187-98. doi: 10.1634/theoncologist.8-2-187. PMID 12697943
- [Result] Vargas-Alarcon G, Ramirez-Bello J, de la Pena A, Calderon-Cruz B, Pena-Duque MA, Martinez-Rios MA, Ramirez-Fuentes S, Perez-Mendez O, Fragoso JM. Distribution of ABCB1, CYP3A5, CYP2C19, and P2RY12 gene polymorphisms in a Mexican Mestizos population. Mol Biol Rep. 2014 Oct;41(10):7023-9. doi: 10.1007/s11033-014-3590-y. Epub 2014 Aug 9. PMID 25106522
- [Result] Kimchi-Sarfaty C, Marple AH, Shinar S, Kimchi AM, Scavo D, Roma MI, Kim IW, Jones A, Arora M, Gribar J, Gurwitz D, Gottesman MM. Ethnicity-related polymorphisms and haplotypes in the human ABCB1 gene. Pharmacogenomics. 2007 Jan;8(1):29-39. doi: 10.2217/14622416.8.1.29. PMID 17187507
- [Result] Siddiqui A, Kerb R, Weale ME, Brinkmann U, Smith A, Goldstein DB, Wood NW, Sisodiya SM. Association of multidrug resistance in epilepsy with a polymorphism in the drug-transporter gene ABCB1. N Engl J Med. 2003 Apr 10;348(15):1442-8. doi: 10.1056/NEJMoa021986. PMID 12686700
- [Result] Tsuji D, Kim YI, Nakamichi H, Daimon T, Suwa K, Iwabe Y, Hayashi H, Inoue K, Yoshida M, Itoh K. Association of ABCB1 polymorphisms with the antiemetic efficacy of granisetron plus dexamethasone in breast cancer patients. Drug Metab Pharmacokinet. 2013;28(4):299-304. doi: 10.2133/dmpk.dmpk-12-rg-084. Epub 2013 Jan 29. PMID 23358260
- [Result] He H, Yin JY, Xu YJ, Li X, Zhang Y, Liu ZG, Zhou F, Zhai M, Li Y, Li XP, Wang Y, Zhou HH, Liu ZQ. Association of ABCB1 polymorphisms with the efficacy of ondansetron in chemotherapy-induced nausea and vomiting. Clin Ther. 2014 Aug 1;36(8):1242-1252.e2. doi: 10.1016/j.clinthera.2014.06.016. Epub 2014 Jul 8. PMID 25012726
- [Result] al-Idrissi HY, Ibrahim EM, Abdullah KA, Ababtain WA, Boukhary HA, Macaulay HM. Antiemetic efficacy of high-dose dexamethasone: randomized, double-blind, crossover study with a combination of dexamethasone, metoclopramide and diphenhydramine. Br J Cancer. 1988 Mar;57(3):308-12. doi: 10.1038/bjc.1988.68. PMID 3281702
- [Result] Ondansetron + dexamethasone vs metoclopramide + dexamethasone + diphenhydramine in prevention of cisplatin-induced emesis. Italian Group For Antiemetic Research. Lancet. 1992 Jul 11;340(8811):96-9. PMID 1352024
- [Result] Prevention of chemotherapy- and radiotherapy-induced emesis: results of Perugia Consensus Conference. Antiemetic Subcommittee of the Multinational Association of Supportive Care in Cancer (MASCC). Ann Oncol. 1998 Aug;9(8):811-9. PMID 9789602
- [Result] Abali H, Celik I. Tropisetron, ondansetron, and granisetron for control of chemotherapy-induced emesis in Turkish cancer patients: a comparison of efficacy, side-effect profile, and cost. Cancer Invest. 2007 Apr-May;25(3):135-9. doi: 10.1080/07357900701208709. PMID 17530482
- [Result] Aapro MS, Grunberg SM, Manikhas GM, Olivares G, Suarez T, Tjulandin SA, Bertoli LF, Yunus F, Morrica B, Lordick F, Macciocchi A. A phase III, double-blind, randomized trial of palonosetron compared with ondansetron in preventing chemotherapy-induced nausea and vomiting following highly emetogenic chemotherapy. Ann Oncol. 2006 Sep;17(9):1441-9. doi: 10.1093/annonc/mdl137. Epub 2006 Jun 9. PMID 16766588
- [Result] Grunberg SM, Dugan M, Muss H, Wood M, Burdette-Radoux S, Weisberg T, Siebel M. Effectiveness of a single-day three-drug regimen of dexamethasone, palonosetron, and aprepitant for the prevention of acute and delayed nausea and vomiting caused by moderately emetogenic chemotherapy. Support Care Cancer. 2009 May;17(5):589-94. doi: 10.1007/s00520-008-0535-9. Epub 2008 Nov 27. PMID 19037667
- [Result] Mustian KM, Darling TV, Janelsins MC, Jean-Pierre P, Roscoe JA, Morrow GR. Chemotherapy-Induced Nausea and Vomiting. US Oncol. 2008;4(1):19-23. doi: 10.17925/ohr.2008.04.1.19. PMID 24761161